CLINICAL TRIAL: NCT06806878
Title: The Effect of Progressive Muscle Relaxation Exercıses Applied to Nursing Students on Success and Anxiety Related to Intramuscular Injection Practice
Brief Title: Progressive Muscle Relaxation Exercises and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Gulden Basit, Assoc. Prof., Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 23841101020
Record Dates: First submitted 2025-01-21; First posted 2025-02-04 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Anxiety State; Progressive Muscle Relaxation; Nursing Students
MeSH Terms: conditions — Anxiety Disorders | interventions — Autogenic Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progressive Muscle Relaxation (Experimental): In this pre-test-post-test randomised controlled study planned to be conducted in Necmettin Erbakan University Faculty of Nursing skills laboratories, consent will be obtained from 1st year nursing students. The students will fill out the descriptive characteristics form, Visual Anxiety Scale and IM injection success test prepared by reviewing the literature before and after intramuscular injection. After the completion of the forms, 'progressive muscle relaxation exercises' will be applied to the students by the researcher for about 30 minutes. Students who volunteered to participate in the study and who took the 'Fundamentals of Nursing' course for the first time will be included in the study.
  Interventions: Other: Progressive muscle relaxation
- no intervention (No Intervention): students will not take any intervention before ım injection application.

INTERVENTIONS:
Other: Progressive muscle relaxation — We will apply progressive muscle relaxation exercises to reduce nursing students' anxiety about intramuscular injection administration
  Arms: Progressive Muscle Relaxation

SUMMARY:
Nursing practice education consists of two parts: laboratory applications aiming at skill acquisition of students and the application part experienced on real patients. Student nurses gain their first skills in laboratory applications accompanied by an instructor. This experience may increase the anxiety levels of nursing students due to reasons such as practising for the first time, hesitating to practice under the supervision of an instructor, and fear of making mistakes. If students learn intramuscular injection, which is one of the skill applications that is a part of care, which is the most important power of nursing, with increased anxiety levels, it may cause a decrease in clinical competence and a decrease in the quality of health care they will provide in the future. Various methods have been tried for nursing students' anxiety levels to be above the optimum level in laboratory applications and it has been observed that anxiety levels have decreased. One of these methods is progressive muscle relaxation exercises. In this study, it is planned to apply progressive muscle relaxation exercises in order to examine the effect of progressive muscle relaxation exercises on the success and anxiety of nursing students related to intramuscular injection practice.

Materials and Method: In this pre-test-post-test randomised controlled study planned to be conducted in Necmettin Erbakan University Faculty of Nursing skill laboratories, consent will be obtained from the 1st year nursing students. The students will fill in the descriptive characteristics form, Visual Anxiety Scale and IM injection success test prepared by reviewing the literature before and after intramuscular injection. After the completion of the forms, 'progressive muscle relaxation exercises' will be applied to the students by the researcher for about 30 minutes. Students who volunteered to participate in the study and who took the 'Fundamentals of Nursing' course for the first time will be included in the study.

DETAILED DESCRIPTION:
In this pre-test-post-test randomised controlled study planned to be conducted in Necmettin Erbakan University Faculty of Nursing skill laboratories, consent will be obtained from the 1st year nursing students. The students will fill in the descriptive characteristics form, Visual Anxiety Scale and IM injection success test prepared by reviewing the literature before and after intramuscular injection. After the completion of the forms, 'progressive muscle relaxation exercises' will be applied to the students by the researcher for about 30 minutes. Students who volunteered to participate in the study and who took the 'Fundamentals of Nursing' course for the first time will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Students who volunteered to participate in the study
* took the 'Fundamentals of Nursing' lesson for the first time

Exclusion Criteria:

* Students who are foreign nationals,
* who have taken the course more than once due to absenteeism or failure,
* who have come with horizontal or vertical transfer,
* who are graduates of Health Vocational High School,
* who have previous injection experience
* who have been diagnosed with anxiety,
* students who do not want to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-03-04 (Actual); Study Completion 2025-03-04 (Actual)

PRIMARY OUTCOMES:
Students anxiety | This scale will be filled out by students before starting the IM injection skill practice and within 10 minutes after the IM practice is completed.
  Students anxiety level will be evaluated by using the "visual anxiety scale" consisting of 100 mm horizontal lines without numbers. At one end of the line is "No Anxiety" and at the other end is "Unbearable Anxiety". The student is expected to put a mark on this line at the point that matches the level of their anxiety. The distance from the lowest level to the student's mark is measured with a ruler and the numerical value of the anxiety level is obtained in cm or mm.

SECONDARY OUTCOMES:
Intramuscular Injection Success Test | this test will be answered before and within 10 minutes after im injection implementation
  Intramuscular Injection Success Test is a test consisting 21 multiple choice question. Each correct answer is considered as "1" point, unanswered questions are not scored. Test scores are evaluated out of a total of 21 points.

CONTACTS AND LOCATIONS:
Overall Officials: Gülden Basit, Dr, Study Chair — Necmettin Erbakan University
Locations (2):
- Turkey (Türkiye) (2):
  - Necmettin Erbakan University, Konya, Meram
  - Necmettin Erbakan University, Meram

IPD SHARING:
Plan to Share IPD: No